CLINICAL TRIAL: NCT01469039
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of ALKS 9072 in Subjects With Acute Exacerbation of Schizophrenia
Brief Title: A Study to Evaluate the Efficacy and Safety of ALKS 9072 (Also Known as Aripiprazole Lauroxil, ALKS 9070, or ARISTADA) in Subjects With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK9072-003
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia
Keywords: Alkermes; schizophrenia; ALKS 9072; ALKS 9070; aripiprazole lauroxil
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALKS 9072 (Experimental)
  Interventions: Drug: ALKS 9072
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 9072 — Intramuscular (IM) injection, 441 mg or 882 mg given monthly
  Arms: ALKS 9072
Drug: Placebo — Placebo for IM injection, given monthly
  Arms: Placebo

SUMMARY:
The study will determine the efficacy of ALKS 9072 (also known as aripiprazole lauroxil or ALKS 9070) for the treatment of schizophrenia in subjects experiencing an acute exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-IV-TR criteria
* Has been able to achieve outpatient status for more than 3 months in the past year
* Body mass index (BMI) of 18.5 to 40.0 kg/m2 (inclusive)
* Resides in a stable living situation
* Willing and able to be confined to an inpatient study unit for 2 weeks or longer

Exclusion Criteria:

* History of poor or inadequate clinical response to treatment with aripiprazole
* History of treatment resistance
* Known or suspected intolerance of, allergy, or hypersensitivity to aripiprazole, its ingredients, other antipsychotic agent, or INTRALIPID (including peanuts, soy, egg, or glycerol)
* Diagnosis of current substance dependence (including alcohol)
* Pregnant, lactating, or breastfeeding
* Receipt of any antipsychotic medication by IM injection within 60 days before Screening
* Current involuntary hospitalization or incarceration
* Hospitalized for more than 30 days during the 90 days before Screening

Additional inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (80):
- United States (23):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Springdale, Arkansas
  - Alkermes Investigational Site, Cerritos, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, La Habra, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Fort Lauderdale, Florida
  - Alkermes Investigational site, Leesburg, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, Overland Park, Kansas
  - Alkermes Investigational Site, Rockville, Maryland
  - Alkermes Investigational Site, Creve Coeur, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Charleston, South Carolina
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Dallas, Texas
- Bulgaria (13):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Kazanlak
  - Alkermes Investigational Site, Novi Iskar
  - Alkermes Investigational Site, Pazardzhik
  - Alkermes Investigational Site, Pleven
  - Alkermes Investigational Site, Plovdiv
  - Alkermes Investigational Site, Radnevo
  - Alkermes Investigational Site, Rousse
  - Alkermes Investigational Site, Sofia
  - Alkermes Investigational Site, Stara Zagora
  - Alkermes Investigational Site, Targovishte
  - Alkermes Investigational Site, Veliko Tarnovo
  - Alkermes Investigational Site, Vratsa
- Malaysia (4):
  - Alkermes Investigational Site, Cheras
  - Alkermes Investigational Site, Johor Bahru
  - Alkermes Investigational Site, Kuala Lumpur
  - Alkermes Investigational Site, Kuching
- Philippines (6):
  - Alkermes Investigational Site, Mariveles, Bataan
  - Alkermes Investigational Site, Cebu City
  - Alkermes Investigational Site, Iloilo City
  - Alkermes Investigational Site, Mandaluyong
  - Alkermes Investigational Site, Manila
  - Alkermes Investigational Site, Pasig
- Romania (5):
  - Alkermes Investigational Site, Oradea, Bihor County
  - Alkermes Investigational Site, Bucharest
  - Alkermes Investigational Site, Craiova
  - Alkermes Investigational Site, Iași
  - Alkermes Investigational Site, Târgu Mureş
- Russia (14):
  - Alkermes Investigational Site, Nikol’skoye, Gatchinckiy
  - Alkermes Investigational Site, Staritsa, Orenburg Oblast
  - Alkermes Investigational Site, Talagi, Primorskiy (Maritime) Kray
  - Alkermes Investigational Site, Khot'kovo, Sergievo-Posadskiy
  - Alkermes Investigational Site, Lipetsk
  - Alkermes Investigational Site, Moscow
  - Alkermes Investigational Site, Nizhny Novgorod
  - Alkermes Investigational Site, Rostov-on-Don
  - Alkermes Investigational Site, Saint Petersburg
  - Alkermes Investigational Site, Samara
  - Alkermes Investigational Site, Saratov
  - Alkermes Investigational Site, Stavropol
  - Alkermes Investigational Site, Voronezh
  - Alkermes Investigational Site, Yaroslavl
- South Korea (3):
  - Alkermes Investigational Site, Jeju City
  - Alkermes Investigational Site, Jeollanam-do
  - Alkermes Investigational Site, Seoul
- Ukraine (12):
  - Alkermes Investigational Site, Stepanivka, Kherson Oblast
  - Alkermes Investigational Site, Chernihiv
  - Alkermes Investigational Site, Donetsk
  - Alkermes Investigational Site, Kharkiv
  - Alkermes Investigational Site, Kyiv
  - Alkermes Investigational Site, Luhansk
  - Alkermes Investigational Site, Lviv
  - Alkermes Investigational Site, Poltava
  - Alkermes Investigational Site, Simferopol
  - Alkermes Investigational Site, Ternopil
  - Alkermes Investigational Site, Uzhhorod
  - Alkermes Investigational Site, Vinnytsia

REFERENCES:
- [Result] Targum SD, Risinger R, Du Y, Pendergrass JC, Jamal HH, Silverman BL. Effect of patient age on treatment response in a study of the acute exacerbation of psychosis in schizophrenia. Schizophr Res. 2017 Jan;179:64-69. doi: 10.1016/j.schres.2016.09.034. Epub 2016 Oct 1. PMID 27707530
- [Result] Nasrallah HA, Newcomer JW, Risinger R, Du Y, Zummo J, Bose A, Stankovic S, Silverman BL, Ehrich EW. Effect of Aripiprazole Lauroxil on Metabolic and Endocrine Profiles and Related Safety Considerations Among Patients With Acute Schizophrenia. J Clin Psychiatry. 2016 Nov;77(11):1519-1525. doi: 10.4088/JCP.15m10467. PMID 27574838
- [Result] Citrome L, Du Y, Risinger R, Stankovic S, Claxton A, Zummo J, Bose A, Silverman BL, Ehrich EW. Effect of aripiprazole lauroxil on agitation and hostility in patients with schizophrenia. Int Clin Psychopharmacol. 2016 Mar;31(2):69-75. doi: 10.1097/YIC.0000000000000106. PMID 26517202
- [Result] Meltzer HY, Risinger R, Nasrallah HA, Du Y, Zummo J, Corey L, Bose A, Stankovic S, Silverman BL, Ehrich EW. A randomized, double-blind, placebo-controlled trial of aripiprazole lauroxil in acute exacerbation of schizophrenia. J Clin Psychiatry. 2015 Aug;76(8):1085-90. doi: 10.4088/JCP.14m09741. PMID 26114240
- [Result] Potkin SG, Risinger R, Du Y, Zummo J, Bose A, Silverman B, Stankovic S, Ehrich E. Efficacy and safety of aripiprazole lauroxil in schizophrenic patients presenting with severe psychotic symptoms during an acute exacerbation. Schizophr Res. 2017 Dec;190:115-120. doi: 10.1016/j.schres.2017.03.003. Epub 2017 Mar 23. PMID 28342578
- [Result] Cameron C, Zummo J, Desai DN, Drake C, Hutton B, Kotb A, Weiden PJ. Aripiprazole Lauroxil Compared with Paliperidone Palmitate in Patients with Schizophrenia: An Indirect Treatment Comparison. Value Health. 2017 Jul-Aug;20(7):876-885. doi: 10.1016/j.jval.2017.03.010. Epub 2017 May 9. PMID 28712616
- [Result] Citrome L, Risinger R, Cutler AJ, Du Y, Zummo J, Nasrallah HA, Silverman BL. Effect of aripiprazole lauroxil in patients with acute schizophrenia as assessed by the Positive and Negative Syndrome Scale-supportive analyses from a Phase 3 study. CNS Spectr. 2018 Aug;23(4):284-290. doi: 10.1017/S1092852917000396. Epub 2017 Jun 19. PMID 28625204
- [Result] Hard ML, Mills RJ, Sadler BM, Turncliff RZ, Citrome L. Aripiprazole Lauroxil: Pharmacokinetic Profile of This Long-Acting Injectable Antipsychotic in Persons With Schizophrenia. J Clin Psychopharmacol. 2017 Jun;37(3):289-295. doi: 10.1097/JCP.0000000000000691. PMID 28350572
- [Result] Cameron C, Zummo J, Desai D, Drake C, Hutton B, Kotb A, Weiden PJ. Efficacy and safety of aripiprazole lauroxil once-monthly versus aripiprazole once-monthly long-acting injectable formulations in patients with acute symptoms of schizophrenia: an indirect comparison of two double-blind placebo-controlled studies. Curr Med Res Opin. 2018 Apr;34(4):725-733. doi: 10.1080/03007995.2017.1410471. Epub 2018 Jan 10. PMID 29179595
- [Derived] Sommi RW, Saklad SR, Weiden PJ, Still D, Wang M, Yagoda S. Initiating Aripiprazole Lauroxil: Post Hoc Analysis of Safety and Tolerability of 1-Day and 21-Day Regimens. J Clin Psychiatry. 2024 Aug 12;85(3):23m15132. doi: 10.4088/JCP.23m15132. PMID 39145678
- [Derived] McEvoy JP, Risinger R, Mykhnyak S, Du Y, Liu CC, Stanford AD, Weiden PJ. Durability of Therapeutic Response With Long-Term Aripiprazole Lauroxil Treatment Following Successful Resolution of an Acute Episode of Schizophrenia. J Clin Psychiatry. 2017 Sep-Oct;78(8):1103-1109. doi: 10.4088/JCP.17m11625. PMID 28937706
- See also: Russian clinical trials website — http://grls.rosminzdrav.ru
- See also: EU Clinical Trials Register; EudraCT number 2012-003445-15 — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Included subjects with schizophrenia experiencing an acute exacerbation episode.
Pre-assignment Details: Subjects were admitted to an inpatient study unit. Currently prescribed antipsychotics were discontinued prior to administration of study drug. One randomized subject was discontinued for a protocol violation prior to receiving investigational treatment.
Groups:
- Aripiprazole Lauroxil 441 mg; Aripiprazole Lauroxil 882 mg; Placebo: Intramuscular injection, given monthly
Period: Overall Study
Arm/Group | Aripiprazole Lauroxil 441 mg | Aripiprazole Lauroxil 882 mg | Placebo
Started | 207 | 208 | 208
Completed | 130 | 135 | 95
Not Completed | 77 | 73 | 113

BASELINE CHARACTERISTICS:
Population: Randomized Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole Lauroxil 441 mg | Aripiprazole Lauroxil 882 mg | Placebo | Total
Number analyzed (Participants) | 207 | 208 | 208 | 623
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 1 | 3
  Between 18 and 65 years | 205 | 207 | 206 | 618
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (10.13) | 39.7 (11.06) | 39.5 (11.85) | 39.7 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 65 | 69 | 200
  Male | 141 | 143 | 139 | 423
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 24 | 28 | 29 | 81
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 83 | 81 | 84 | 248
  White | 99 | 98 | 94 | 291
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 103 | 102 | 102 | 307
  Philippines | 16 | 21 | 16 | 53
  Malaysia | 7 | 7 | 10 | 24
  Ukraine | 29 | 29 | 32 | 90
  Romania | 5 | 6 | 6 | 17
  Bulgaria | 23 | 19 | 17 | 59
  Russian Federation | 24 | 24 | 25 | 73

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline at Day 85 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS scale contains 30 questions, each containing an answer range of 1-7. A total PANSS score can range from between 30 to 210; a higher score indicates a worse disease condition.
Time Frame: Data collected from baseline to day 85
Population: Full Analysis Set (FAS) defined as all randomized subjects who received at least 1 dose of IM study drug and had at least 1 primary efficacy assessment after administration of IM study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil 441 mg | Aripiprazole Lauroxil 882 mg | Placebo
Number analyzed (Participants) | 196 | 204 | 196
units on a scale | -20.9 (1.39) | -21.8 (1.35) | -9.8 (1.39)
Statistical Analysis 1: Comparison: Aripiprazole Lauroxil 441 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Aripiprazole Lauroxil 882 mg; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Scores at Day 85
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the study. Results indicate participants evaluated at one of the following categories: "1: very much improved"; "2: much improved"; "3: minimally improved"; "4: no change"; "5: minimally worse"; "6: much worse"; or "7: very much worse".
Time Frame: 85 Days
Population: FAS, defined as all randomized subjects who received at least 1 IM dose of study drug and had at least 1 primary efficacy assessment after administration of IM study drug.
Measure: Number; unit: participants in category
Arm/Group | Aripiprazole Lauroxil 441 mg | Aripiprazole Lauroxil 882 mg | Placebo
Number analyzed (Participants) | 196 | 204 | 196
participants in category
  CGI Score: Very much improved | 27 | 25 | 15
  CGI Score: Much improved | 68 | 81 | 33
  GCI Score: Minimally improved | 45 | 52 | 43
  CGI Score: No change | 32 | 24 | 42
  CGI Score: Minimally worse | 11 | 16 | 37
  CGI Score: Much worse | 12 | 5 | 23
  CGI Score: Very much worse | 1 | 1 | 3
Statistical Analysis 1: Comparison: Aripiprazole Lauroxil 441 mg; Test type: Superiority or Other; p < 0.001, Wilcoxon rank sum test based on LOCF — significant p-value, active vs placebo
Statistical Analysis 2: Comparison: Aripiprazole Lauroxil 882 mg; Test type: Superiority or Other; p < 0.001, Wilcoxon rank sum test based on LOCF — significant p-value, active vs placebo

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 85-day treatment period.
Description: One randomized subject was discontinued for a protocol violation prior to receiving IM study drug (placebo), and this subject was not included in the safety population. This changes the overall number of subjects in the placebo group to include 207.
Arm/Group | Aripiprazole Lauroxil 441 mg | Aripiprazole Lauroxil 882 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/207 | 4/208 | 4/207
Other Adverse Events (participants affected / at risk) | 66/207 | 68/208 | 76/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole Lauroxil 441 mg (N=207) | Aripiprazole Lauroxil 882 mg (N=208) | Placebo (N=207)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug Abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Victim of homicide (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole Lauroxil 441 mg (N=207) | Aripiprazole Lauroxil 882 mg (N=208) | Placebo (N=207)
Akathisia (Nervous system disorders) | 24 (26) | 23 (30) | 9 (9)
Headache (Nervous system disorders) | 17 (20) | 18 (22) | 17 (20)
Agitation (Psychiatric disorders) | 3 (4) | 3 (3) | 11 (11)
Anxiety (Psychiatric disorders) | 6 (11) | 11 (14) | 14 (16)
Insomnia (Psychiatric disorders) | 20 (26) | 25 (27) | 24 (29)
Schizophrenia (Psychiatric disorders) | 12 (13) | 5 (5) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.